CLINICAL TRIAL: NCT02527629
Title: Aortic Replacement Using Individualised Regenerative Allografts: Bridging the Therapeutic Gap - ARISE (the "Surveillance")
Brief Title: Aortic Replacement Using Individualised Regenerative Allografts - ARISE (the "Surveillance")
Acronym: ARISE
Status: Completed | Type: Observational
Sponsor: corlife (Industry)
Collaborators: Hannover Medical School (Other); Leiden University Medical Center (Other); Azienda Ospedaliera di Padova (Other); Hospital Clinic of Barcelona (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Universitaire Ziekenhuizen KU Leuven (Other); Heinrich-Heine University, Duesseldorf (Other); Vienna General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015- 01, 20.07.2015; Grant Agreement No: 643597 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2015-07-27; First posted 2015-08-19 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Heart Valve Disease
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Decellularized human valves: Aortic heart valve replacement
  Interventions: Other: Decellularized human heart valves

INTERVENTIONS:
Other: Decellularized human heart valves — Decellularized human aortic heart valves
  Other Names: Arise Aortic Valve (AV)

SUMMARY:
Evaluation of decellularized human heart valves for aortic heart valve replacement in comparison to current valve substitutes.

Safety endpoints include cardiovascular adverse events, time to re-operation, re-intervention and explantation.

Efficacy endpoints include freedom from valve dysfunction and hemodynamic performance.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single-arm, multi-centre surveillance study to be conducted in Europe.

The Surveillance is designed as a study, where

* ARISE AV is prescribed in the usual manner in accordance with the terms of the approval.
* Assignment of the patient to a particular therapeutic strategy is not decided in advance by this Surveillance Protocol but falls within current practice and the prescription of ARISE AV is clearly separated from the decision to include the patient in the Surveillance.
* No additional diagnostic or monitoring procedures shall be applied to the patients.
* and epidemiological methods shall be used for the analysis of collected data.

ELIGIBILITY:
Inclusion Criteria:

i. Indication for aortic valve replacement according to current medical guidelines in valvular heart disease

ii. Informed consent of legal guardians or patients, assent of patients

Exclusion Criteria:

i. The patient has not provided Surveillance informed consent.

ii. The patient shall not suffer from:

* generalized connective tissue disorders (eg, Marfan syndrome), or .
* active rheumatic disorders, or
* severe asymmetric calcification of the valve ring.

iii. The coronary arteries of the patient shall not be in abnormal position or heavily calcified.

iv. Patients shall not show hypersensitivity against sodium dodecyl sulphate (SDS), sodium desoxycholate (SDC), human collagen (or other elastic fibers) or Benzonase®.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe aortic valve disease and the indication for aortic valve replacement
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2015-09; Primary Completion 2019-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Adverse Reactions (AR) | up to 24 months
  Rate of cardiovascular AR, e.g. all-cause mortality, major stroke, life-threatening (or disabling) bleeding, acute kidney injury-stage 3 (including renal replacement therapy), peri-procedural myocardial infarction, major vascular complication, repeat procedure for valve-related dysfunction (surgical or interventional therapy).
Freedom from valve dysfunction at end of the study | up to 24 months
  Echocardiographic studies should be obtained and analyzed at discharge and at 3, 6 Months and at annual follow-ups. The requested variables include peak and mean systolic gradient, using pw and cw doppler, in the left ventricular outflow tract, respective the aortic valve. The echo evaluation (videotape or CD) should remain at the Surveillance site, but be available to corlife Surveillance personnel upon request. The MRIs will be analyzed by the MRI Core Laboratory at Medical School in Hannover for potential valvular stenosis, via phase contrast flow measurements in the aorta and for valvular competence, via phase contrast flow measurements and by ventricular volumetry. MRI cine images will be used to visualize the Surveillance valve in patients with poor echocardiographic windows.

SECONDARY OUTCOMES:
Evaluation of composite blood parameters | up to 24 months
  The following data should be collected: Hb, LDH, Haptoglobin, CRP, Leukocytes. Blood studies should be performed within 7 days preoperatively and at discharge. Blood data will support the absence/presence of related AR. For example, haemolysis should be reported as an adverse event if anaemia is present; however, in the absence of anaemia, haemolysis will be considered to be compensated and does not require reporting. Time to events, such as death, reoperation including explantation will be evaluated for those outcomes, calculated from the date of operation.
Time to reoperation and / or death | up to 24 months
  Time to events, such as death, reoperation including explantation will be evaluated for those outcomes, calculated from the date of operation
Evaluation of composite valve measures | up to 24 months
  Diameters of ARISE AV at end of the Surveillance will be analyzed in comparison to diameters at implantation and to age matched reference values. Preoperative non-invasive data on left ventricular size and function, such as left ventricular end diastolic, end systolic volume, ejection fraction and ventricular mass will be derived from MRI and compared to postoperative status.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Haverich, Prof. Dr., Principal Investigator — Hannover Medical School; Samir Sarikouch, PD Dr., Study Director — Hannover Medical School
Locations (8):
- Universitair Ziekenhuis Leuven, UZL, Leuven, Belgium
- Germany (2):
  - University of Düsseldorf, Department of Cardiovascular Surgery, Düsseldorf
  - Hannover Medical School, Hanover
- Azienda Ospedaliera di Padova, U.O.C. di Cardiochirurgia Pediatrica e Cardiopatie Congenite, Padua, Italy
- Leids Universitair Medisch Centrum, LUMC, Leiden, Netherlands
- University Hospital Clinic de Barcelona, Cardiovascular Surgery administrative area, Barcelona, Spain
- Kinderspital Zürich, Zurich, Switzerland
- Royal Brompton and Harefield National Health Service Trust, London, United Kingdom

REFERENCES:
- [Result] Horke A, Tudorache I, Laufer G, Andreas M, Pomar JL, Pereda D, Quintana E, Sitges M, Meyns B, Rega F, Hazekamp M, Hubler M, Schmiady M, Pepper J, Rosendahl U, Lichtenberg A, Akhyari P, Jashari R, Boethig D, Bobylev D, Avsar M, Cebotari S, Haverich A, Sarikouch S. Early results from a prospective, single-arm European trial on decellularized allografts for aortic valve replacement: the ARISE study and ARISE Registry data. Eur J Cardiothorac Surg. 2020 Nov 1;58(5):1045-1053. doi: 10.1093/ejcts/ezaa100. PMID 32386409
- [Derived] Cvitkovic T, Horke A, Bobylev D, Avsar M, Holst T, Beerbaum P, Boethig D, Petena E, Tsimashok V, Westhoff-Bleck M, Gutberlet M, Beyer FH, Wacker F, Ruhparwar A, Vogel-Claussen J, Sarikouch S, Czerner C. Aortic Compliance After Root Replacement With Decellularized Homografts Versus in Donor Age-Matched Healthy Controls. Interdiscip Cardiovasc Thorac Surg. 2026 Jan 6;41(1):ivaf303. doi: 10.1093/icvts/ivaf303. PMID 41467751
- Available data/document: Study results — https://pubmed.ncbi.nlm.nih.gov/32386409/